CLINICAL TRIAL: NCT05856396
Title: Maternal Determinants of Infant Immunity to Pertussis
Acronym: MADI-02
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Saint Pierre (Other)
Collaborators: Université Libre de Bruxelles (Other)
Responsible Party: Principal Investigator, Tessa Goetghebuer, Head of Clinic, Centre Hospitalier Universitaire Saint Pierre
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: B0762022220909
Record Dates: First submitted 2022-10-05; First posted 2023-05-12 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Vaccination; Infection; Maternal-Fetal Relations; Pertussis; Immunoglobulins
MeSH Terms: conditions — Infections; Whooping Cough | interventions — adacel; Vaxelis

STUDY DESIGN:
Intervention Model Description: * Non pregnant and pregnant women will be recruited in parallel
  * Infants born to Tdap vaccinated-mothers (enrolled or not in the study) or not vaccinated mothers will be recruited
Who Masked: Outcomes Assessor
Masking Description: Researchers analyzing the immunological outcomes will be blinded to the groups of the subjects (pregnant vs non pregnant ; infants)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Pregnant women (Active Comparator): Pregnant women will receive one dose of Pertussis-containing vaccine during pregnancy.
  Interventions: Biological: Triaxis® (Pertussis-containing vaccine)
- Non pregnant women (Active Comparator): Non-Pregnant women will receive one dose of Pertussis-containing vaccine.
  Interventions: Biological: Triaxis® (Pertussis-containing vaccine)
- Infants born to Tdap-vaccinated mothers (Active Comparator): Infants whose mothers have been immunized during pregnancy with Tdap vaccine. Infants will receive three doses of Pertussis-containing vaccine (with 28 days interval starting at two months of age).
  Interventions: Biological: Vaxelis® (Pertussis-containing vaccine)
- Infants born to non Tdap-vaccinated mothers (Active Comparator): Infants whose mothers have not been immunized during pregnancy with Tdap vaccine.
  Infants will receive three doses of Pertussis-containing vaccine (with 28 days interval starting at two months of age).
  Interventions: Biological: Vaxelis® (Pertussis-containing vaccine)

INTERVENTIONS:
Biological: Triaxis® (Pertussis-containing vaccine) — Triaxis® (Pertussis-containing vaccine) will be administered:
  * in non-pregnant women presenting to the Travel and Vaccine clinic for pertussis immunization only or hospital member staff requiring Tetanus Toxoid (TT)-booster immunisation
  * in Pregnant women between 16 and 29 weeks of gestation.
  Arms: Non pregnant women; Pregnant women
Biological: Vaxelis® (Pertussis-containing vaccine) — Vaxelis® (Hexavalent vaccine) will be proposed in infants at 8, 12 and 16 weeks of life.
  Arms: Infants born to Tdap-vaccinated mothers; Infants born to non Tdap-vaccinated mothers

SUMMARY:
The overall objective of the project is to identify the determinants of antibody-mediated immunity in infants born to mothers immunized during pregnancy. Using maternal pertussis immunization as a model, the project will identify key predictors and potential determinants of vaccine responses in pregnant women, of the transfer of maternal antibodies to the newborn and of vaccine responses in infants. A systems biology approach will be used to delineate pre-vaccination and post-vaccination cellular and molecular correlates of the immune response to pertussis immunization in peripheral blood and in breastmilk.

DETAILED DESCRIPTION:
The overall objective of the project is to identify the determinants of antibody-mediated immunity to pertussis in infants born to mothers immunized during pregnancy. Three specific objectives will be targeted:

1. Determine the impact of pregnancy on the quality of antibody response to pertussis immunization and identify immune predictors of vaccine responses in pregnant and non-pregnant women.
2. Identify immune predictors of the transfer of maternal antibodies to the newborn and the presence of antibody in breastmilk following pertussis immunization during pregnancy.
3. Determine the impact of maternal antibodies on the quality of antibody response to pertussis immunization in infants born to mothers immunized or not immunized during pregnancy and identify immune predictors of vaccine responses in the first months of life.

To reach these objectives, 40 non-pregnant and 80 pregnant women will be recruited into the study and vaccinated with a single dose of a pertussis containing vaccine (Triaxis). Blood samples will be collected from:

* non-pregnant women: before vaccination, and day 1/7/28 and month 5 post-vaccination.
* pregnant women: before vaccination, day 1/7/28 post-vaccination, at delivery, and week 6/12 post-delivery. At week 6/12 post-delivery, breast milk samples will be collected as well.

At delivery, a placenta fragment will be collected.

In addition, infants 2-3 months old born either from mothers who were not vaccinated against pertussis during pregnancy (n=40) or born from mothers who were vaccinated against pertussis during pregnancy (n=80) will be recruited in the study. Infants will be vaccinated with three doses of a pertussis containing vaccine (Vaxelis), each one month apart starting from 2-3 months of age. Blood samples will be collected from:

* infants from vaccinated mothers: cord blood, before 1st vaccine dose, day 1 post 1st vaccine dose, before 3rd vaccine dose, and day 28 post 3rd vaccine dose.
* infants from unvaccinated mothers: before 1st vaccine dose, day 1 post 1st vaccine dose, before 3rd vaccine dose, and day 28 post 3rd vaccine dose.

ELIGIBILITY:
Inclusion Criteria:

* For non-pregnant & pregnant women Age between 18 and 45 years Eligible for Tdap vaccination
* For infants Born to mothers vaccinated or not with Tdap Vaccinated with hexavalent vaccine Age between 2 and 3 months

Exclusion Criteria:

* For pregnant and non-pregnant women

  * Inability to understand the nature and extent of the study and the procedures required
  * Grade III/IV anemia,
  * Acute infection at the time of immunization
  * Chronic infections such as Hepatitis B Virus (HBV), Hepatitis C Virus (HCV) or Human Immunodeficiency Virus (HIV) infection, acute toxoplasmosis
  * Current or recent use of immunosuppressive drugs
  * Active neoplasia
  * Other vaccine(s) administered at the same time as Tdap vaccination (wash out of 4 weeks after others vaccinations and 28 days after Tdap vaccination )
* For pregnant women

  * Risk of premature delivery or intrauterine growth retardation
  * Twin or triplet pregnancies
* For non-pregnant women Last Tdap vaccination < 12 months before

For infants:

* Infants born before 35 weeks of gestation
* Birthweight below 2.5 kg,
* Severe neonatal distress
* Serious congenital abnormalities or congenital infection.

Ages: 2 Months to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 200 (Actual)
Dates: Start 2023-09-12 (Actual); Primary Completion 2025-12-23 (Actual); Study Completion 2025-12-23 (Actual)

PRIMARY OUTCOMES:
IgG titers specific to Bordetella Pertussis Antigens by Enzyme-linked immunosorbent assay (ELISA) | Day 28 post-vaccination
  IgG titers specific to Bordetella Pertussis Antigens will be assessed by ELISA:
  * in women (pregnant and non-pregnant) at 28 days post vaccination
  * in infants (from unvaccinated mothers and mothers vaccinated during pregnancy) at 28 days post third vaccine dose
IgG titers specific to Bordetella Pertussis Antigens by Enzyme-linked immunosorbent assay (ELISA) | At delivery
  IgG titers specific to Bordetella Pertussis Antigens will be assessed by ELISA:
  * in women vaccinated during pregnancy, at delivery
  * in umbilical cord blood of infants born to mothers vaccinated during pregnancy

SECONDARY OUTCOMES:
IgG titers specific to Bordetella Pertussis Antigens by Enzyme-linked immunosorbent assay (ELISA) | up to 9 month after vaccination
  IgG titers specific to Bordetella Pertussis Antigens will be assessed by ELISA:
  * in pregnant women (PW): at day of vaccination , day 7 post-vaccination, week 6 and 12 post-delivery
  * in non-pregnant women (non PW): at day of vaccination, day 7 and Month 5 post-vaccination
  * in infants (from unvaccinated mothers and mothers vaccinated during pregnancy) at day of first and third vaccine dose
CD4+ T cell frequencies specific to Bordetella Pertussis Antigens by flow cytometry | up to 9 month after vaccination
  The percentage of CD4+ T cells expressing any of the following biomarkers (CD154, Interferon gamma, IL-2) in response to in vitro stimulation with Bordetella Pertussis Antigens will be measured by flow cytometry:
  i. in pregnant and non-pregnant women: at day of vaccination, and day 28 post vaccination
  ii. in infants (from unvaccinated mothers and mothers vaccinated during pregnancy) at day of first vaccine dose and 28 days after third vaccine dose

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Saint-Pierre, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF

REFERENCES:
- [Background] Marchant A, Sadarangani M, Garand M, Dauby N, Verhasselt V, Pereira L, Bjornson G, Jones CE, Halperin SA, Edwards KM, Heath P, Openshaw PJ, Scheifele DW, Kollmann TR. Maternal immunisation: collaborating with mother nature. Lancet Infect Dis. 2017 Jul;17(7):e197-e208. doi: 10.1016/S1473-3099(17)30229-3. Epub 2017 Apr 19. PMID 28433705
- [Background] Gunn BM, Alter G. Modulating Antibody Functionality in Infectious Disease and Vaccination. Trends Mol Med. 2016 Nov;22(11):969-982. doi: 10.1016/j.molmed.2016.09.002. Epub 2016 Oct 15. PMID 27756530
- [Background] Jennewein MF, Alter G. The Immunoregulatory Roles of Antibody Glycosylation. Trends Immunol. 2017 May;38(5):358-372. doi: 10.1016/j.it.2017.02.004. Epub 2017 Apr 3. PMID 28385520
- [Background] Jennewein MF, Abu-Raya B, Jiang Y, Alter G, Marchant A. Transfer of maternal immunity and programming of the newborn immune system. Semin Immunopathol. 2017 Nov;39(6):605-613. doi: 10.1007/s00281-017-0653-x. Epub 2017 Oct 2. PMID 28971246
- [Background] Jennewein MF, Goldfarb I, Dolatshahi S, Cosgrove C, Noelette FJ, Krykbaeva M, Das J, Sarkar A, Gorman MJ, Fischinger S, Boudreau CM, Brown J, Cooperrider JH, Aneja J, Suscovich TJ, Graham BS, Lauer GM, Goetghebuer T, Marchant A, Lauffenburger D, Kim AY, Riley LE, Alter G. Fc Glycan-Mediated Regulation of Placental Antibody Transfer. Cell. 2019 Jun 27;178(1):202-215.e14. doi: 10.1016/j.cell.2019.05.044. Epub 2019 Jun 13. PMID 31204102
- [Background] Jennewein MF, Kosikova M, Noelette FJ, Radvak P, Boudreau CM, Campbell JD, Chen WH, Xie H, Alter G, Pasetti MF. Functional and structural modifications of influenza antibodies during pregnancy. iScience. 2022 Mar 16;25(4):104088. doi: 10.1016/j.isci.2022.104088. eCollection 2022 Apr 15. PMID 35402869
- [Background] Tsang JS. Utilizing population variation, vaccination, and systems biology to study human immunology. Trends Immunol. 2015 Aug;36(8):479-93. doi: 10.1016/j.it.2015.06.005. Epub 2015 Jul 14. PMID 26187853